CLINICAL TRIAL: NCT04811053
Title: A Phase Ⅱ, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of HR021618 in the Treatment of Moderate to Severe Pain After Abdominal Surgery
Brief Title: HR021618 in Moderate to Severe Pain After Abdominal Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR021618-203
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Pain After Abdominal Surgery

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental)
  Interventions: Drug: HR021618
- Treatment group B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HR021618 — Treatment group A: HR021618 injection
  Arms: Treatment group A
Drug: Placebo — Treatment group B: Saline injection
  Arms: Treatment group B

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of HR021618 in the treatment of moderate to severe pain after abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Subjects requiring elective general anesthesia abdominal surgery
3. Male or female
4. Meet BMI standard
5. Conform to the ASA Physical Status Classification

Exclusion Criteria:

1. Subjects with a history of abdominal surgery
2. Subjects had hemorrhagic disorders
3. Subjects had cardiac, serious hepatic or renal, cardiovascular or cerebrovascular, metabolic, psychiatric disorders, chronic pain, or malignant tumors
4. Subjects with poor blood pressure control after medication
5. Abnormal QTc
6. Abnormal random blood glucose
7. Abnormal values in the laboratory
8. Allergic to meloxicam or any excipient of HR021618, aspirin, other non-steroidal anti-inflammatory drugs (NSAIDs) or to any peri- or postoperative medications used in this study
9. Use other drugs that affect the analgesic effect before randomization, and the time from the last use to randomization is shorter than 5 half-lives
10. Pregnant or nursing women
11. No birth control during the specified period of time
12. Participated in clinical trials of other drugs (received experimental drugs)
13. The inestigators determined that other conditions were inappropriate for participation in this clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
AUC48 | 48 hours after recovery from anesthesia] Area under the pain intensity-time curve.
  Area under the pain intensity-time curve.

SECONDARY OUTCOMES:
Total consumption of morphine over 0-48, 0-24, 24-48 hours | 48 hours after recovery from anesthesia
  Total consumption of morphine after recovery from anesthesia.
AUC3, AUC24, AUC15-21, AUC18-24, AUC24-28, AUC39-45, AUC42-48 | 48 hours after recovery from anesthesia
  Area under the pain intensity-time curve.
Time of the first dose of rescue analgesia | 48 hours after recovery from anesthesia
  Time of the first dose of rescue analgesia after recovery from anesthesia.
Proportion of subjects receiving rescue analgesia | 48 hours after recovery from anesthesia
  Proportion of subjects receiving rescue analgesia after recovery from anesthesia.
Frequency of doses of rescue analgesia | 48 hours after recovery from anesthesia
  Frequency of doses of rescue analgesia after recovery from anesthesia.
Subjects' satisfaction rating | 48 hours after recovery from anesthesia
  Subjects' satisfaction rating.
Anesthesiologist satisfaction rating | 48 hours after recovery from anesthesia
  Anesthesiologist satisfaction rating.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China